CLINICAL TRIAL: NCT04125160
Title: Markers for Glycaemic Control and Continuous Glucose Monitoring in Persons With Type 2 Diabetes on Peritoneal Dialysis
Brief Title: Glycaemic Markers in Persons With Type 2 Diabetes on Peritoneal Dialysis
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Zealand University Hospital (Other); Herlev Hospital (Other); Hillerod Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Bo Feldt-Rasmussen, Professor, DMSc, Head of Nephrology, Rigshospitalet, Denmark
Other Study IDs: GLYCO-PD
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: HbA1c; Peritoneal Diseases; Glycated Albumin; Fructosamine; Continuous Glucose Monitoring
MeSH Terms: conditions — Peritoneal Diseases | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Type 2 diabetes and peritoneal dialysis: Case group with type 2 diabetes undergoing peritoneal dialysis for at least 3 months.
  Interventions: Device: Continuous glucose monitoring; Diagnostic Test: Glycaemic markers
- Type 2 diabetes and eGFR above 60ml/min: Control group with type 2 diabetes and no nephropathy (defined as eGFR above 60ml/min and UACR below 300mg/g).
  Interventions: Device: Continuous glucose monitoring; Diagnostic Test: Glycaemic markers

INTERVENTIONS:
Device: Continuous glucose monitoring — Continuous glucose monitoring over 16 days
Diagnostic Test: Glycaemic markers — Measurement of HbA1c, glycated albumin and fructosamine.

SUMMARY:
The aim is to investigate the correlation between mean glucose measured by continuous glucose monitoring (CGM) and mean glucose estimated from glycated haemoglobin A1c (HbA1c) in persons with type 2 diabetes undergoing peritoneal dialysis compared with patients with type 2 diabetes and normal renal function. Furthermore, the aim is to compare CGM and HbA1c with glycated albumin and fructosamine.

DETAILED DESCRIPTION:
Background:

In persons with type 2 diabetes, glycated haemoglobin A1c (HbA1c) is used as an indirect measure of the mean glucose over the past 3-4 months. The normal range of HbA1c and the correlation to the mean glucose has been determined from studies in subjects without severe chronic kidney disease.

In persons with end-stage renal disease (ESRD) and type 2 diabetes, HbA1c has been shown in small studies to underestimate mean glucose when compared with continuous glucose monitoring (CGM) or alternative glycaemic markers such as glycated albumin or fructosamine. The cause of a falsely low HbA1c in persons with ESRD and diabetes is not clear, but adjuvant erythropoietin treatment and iron infusion increase erythropoiesis, thus increasing the number of new non-glycated erythrocytes that are thought to lower HbA1c. Furthermore, the erythrocyte life span was found to be decreased in individuals receiving hemodialysis and peritoneal dialysis, which may also contribute to a reduction in HbA1c.

CGM is an alternative to HbA1c in glycaemic monitoring and measures interstitial glucose that calibrates with blood glucose within minutes. CGM measures interstitial glucose every five minutes for up to eight days (Medtronic's Ipro2). Studies of persons with type 1 diabetes and CGM measurements performed over three months showed that approximately two-weeks of CGM measurements correlated to HbA1c. When CGM was performed beyond 14 days, the correlation between the mean glucose from CGM and HbA1c improved only modestly.

Values of CGM measurements also provide a basis for monitoring glycaemic variability, time-in-range and hypoglycaemic episodes. For persons with diabetes undergoing peritoneal dialysis, there are only a few studies validating HbA1c and none have been prospective with a control group over a long period of time. A retrospective study of 60 persons with diabetes and in peritoneal dialysis (without control group) found a significant correlation between HbA1c and mean interstitial glucose as measured by CGM (r = 0.48, P≤0.0001). A prospective study of 25 persons with diabetes and in peritoneal dialysis (without control group) also found a significant correlation (r = 0.51, P≤0.01). A study of three persons with diabetes and in peritoneal dialysis (without control group) found that HbA1c compared to CGM underestimated mean glucose in one, but overestimated mean glucose in the other two. However, all three studies did not include a control group and had few days of CGM measurements, which collectively mean that the evidence for the use of HbA1c in this patient group is sparse.

In a study of peritoneal dialysis subjects with diabetic nephropathy (n = 1296), 17.7% had normal HbA1c and were without antidiabetic treatment. When the same study included glycated albumin, 10.9% were found to have normal HbA1c, normal glycated albumin (defined as less than 16%) and were without antidiabetic medication. The study concluded that normal HbA1c alone overestimates the prevalence of burnt-out diabetes.

The uncertainty associated with HbA1c in persons with type 2 diabetes undergoing peritoneal dialysis is a problem both in terms of diagnosing and treating diabetes appropriately. CGM, glycated albumin and fructosamine are independent of erythrocyte turnover thus allowing for a validation of HbA1c in this group of patients.

Objective:

To investigate the correlation between mean glucose measured by continuous glucose monitoring (CGM) and mean glucose estimated from glycated haemoglobin A1c (HbA1c) in persons with type 2 diabetes undergoing peritoneal dialysis compared with a control group of persons with type 2 diabetes and normal renal function.

Method:

Prospective case-control study over 16 days with 26 persons in each group. The case group consist of persons with type 2 diabetes undergoing peritoneal dialysis and the control group consists of persons with type 2 diabetes with normal renal function (defined as an estimated glomerular filtration rate (eGFR) above 60 ml/min and urine albumin-creatinine ratio below 300mg/g). CGM is performed for a maximum of 16 days. On visit 1 (day 0), CGM is performed for 8 days and visit 2 (day 8) (+7/-4 days), CGM is performed for another 8 days. Glycaemic markers are measured at baseline and on visit 3 (final day of the study). At least 12 days of CGM must be completed for each person. Data is collected using REDcap.

Statistics:

The null hypothesis is that there is no difference in the ratio between the two groups measured as mean glucose concentration measured over 16 days at CGM (mmol / L) divided by the estimated glucose concentration from HbA1c (mmol / L) measured at day 16.

The alternative hypothesis is that there is a 17% difference between groups for the ratio of mean glucose concentration measured by CGM (mmol / L) divided by the mean glucose concentration from HbA1c (mmol / L). In a pilot study of persons with type 2 diabetes and dialysis dependent ESRD compared with persons with normal renal function, a 17% difference was found in the ratio between the two groups. In a two-sided unpaired t-test with α = 0.05, SD = 1.17 and power of 90%, a sample size of 24 individuals in each group will show a significant difference. A drop of approximately 10% is expected and a total of 26 are included in each group.

ELIGIBILITY:
Inclusion criteria for case group (on peritoneal dialysis with type 2 diabetes):

* Type 2 diabetes*
* BMI 17.5-50 kg/m2
* Receiving antidiabetic treatment
* Peritoneal dialysis treatment for a minimum of 3 months

Exclusion criteria for case group (on peritoneal dialysis with type 2 diabetes):

* Type 1 diabetes
* Acute or chronic pancreatitis
* Intermittent treatment with steroid during study period (defined as more than two days)
* Haemoglobin < 5.5 mmol / l
* Hypertriglyceridemia (≥ 10mmol / L)
* Hyperbilirubinemia (≥ 35 μmol / L)
* Pregnant or breast-feeding
* Blood transfusion within the last 3 months
* Blood transfusion during the investigation period
* Splenectomy
* High alcohol consumption (defined as more than 21 units per week)
* Vitamin E supplement
* Ribavirin treatment
* Interferon Alpha treatment
* Positive for haemoglobinopathy (examined for haemoglobinopathy if patients come from Africa, Mediterranean, Middle East, Iran, Iraq, India, Pakistan or Southeast Asia)
* Severe infections

Inclusion criteria for control group (type 2 diabetes and normal renal function):

* Type 2 diabetes*
* BMI 17.5-50 kg / m2
* Receiving antidiabetic treatment
* eGFR > 60 ml/min/1.73m2
* Urine Albumin-to-Creatinine Ratio < 300mg/g

Exclusion criteria for control group (type 2 diabetes and normal renal function):

* Type 1 diabetes
* Acute or chronic pancreatitis
* Intermittent treatment with steroid during study period
* Haemoglobin <7.3 mmol / l for women
* Haemoglobin <8.3 mmol / l for men
* Hypertriglyceridemia (≥ 10mmol / L)
* Hyperbilirubinemia (≥ 35 μmol / L)
* Pregnant or breast-feeding
* Blood transfusion within the last 3 months
* Blood transfusion during the investigation period
* Splenectomy
* High alcohol consumption (defined as more than 21 units per week)
* Vitamin E supplement
* Ribavirin
* Interferon Alpha treatment
* Positive for haemoglobinopathy (examined for haemoglobinopathy if patients come from Africa, Mediterranean, Middle East, Iran, Iraq, India, Pakistan or Southeast Asia)
* Severe infections

  *Inclusion with diagnosis of type 2 diabetes was defined as ongoing antidiabetic treatment and previously diagnosed with type 2 diabetes according to the following criteria:
* A random venous plasma glucose concentration ≥ 11.1 mmol/l or
* A fasting plasma glucose concentration ≥ 7.0 mmol/l (whole blood ≥ 6.1 mmol/l) or
* Two hour plasma glucose concentration ≥ 11.1 mmol/l two hours after 75g anhydrous glucose in an oral glucose tolerance test or
* HbA1c above 48 mmol/mol

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Total of 52 participants with 26 in each group.
  Case group: 26 patients on peritoneal dialysis with type 2 diabetes.
  Control group: 26 patients with type 2 diabetes and normal renal function (defined as eGFR >60 ml/min and with Urine Albumin-to-Creatinine Ratio below 300mg/g.
  The patients are recruited from the department of Endocrinology or Nephrology at Rigshospitalet, from Herlev Hospital department of Nephrology, Steno Diabetes Center Copenhagen, Hillerød Hospital department of Nephrology and Roskilde Hospital department of Nephrology.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-09-03 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
HbA1c evaluated by the total mean glucose from continuous glucose monitoring | 16 days
  Difference between the two groups in the ratio of mean glucose measured by continuous glucose monitoring (measured over 16 days) divided by the estimated mean blood glucose from HbA1c (measured at the final visit). For each person at least 12 days of CGM must be completed.

SECONDARY OUTCOMES:
Glycated albumin | 16 days
  Correlation between mean glucose from continuous glucose monitoring (measured over 16 days) and glycated albumin ((%) measured at the final visit).
Fructosamine | 16 days
  Correlation between mean glucose from continuous glucose monitoring (measured over 16 days) and fructosamine ((μmol/l) measured at the final visit).
Standard deviation | 16 days
  Standard deviation for glycaemic variability measured by continuous glucose monitoring in both groups.
Coefficient variation | 16 days
  Coefficient variation for glycaemic variability measured by continuous glucose monitoring in both groups.
Low Blood Glucose Index | 16 days
  Low Blood Glucose Index for glycaemic variability measured by continuous glucose monitoring in both groups. Is a risk index for predicting hypoglycaemia.
High Blood Glucose Index | 16 days
  High Blood Glucose Index for glycaemic variability measured by continuous glucose monitoring in both groups. Is a risk index for predicting hyperglycaemia.
Time in hypoglycaemic range below 3.0 mmol/l | 16 days
  Time in hypoglycaemic range(%) below 3.0 mmol/l evaluated by continuous glucose monitoring .
Time in hypoglycaemic range below 3.9 mmol/l to 3.0 mmol/l | 16 days
  Time in hypoglycaemic range(%) below 3.9 mmol/l to 3.0 mmol/l evaluated by continuous glucose monitoring .
Time in hyperglycaemic range above 10.0 mmol/l | 16 days
  Time in hyperglycaemic range(%) above 10.0 mmol/l evaluated by continuous glucose monitoring .
Time in hyperglycaemic range above 13.9 mmol/l | 16 days
  Time in hyperglycaemic range(%) above 13.9 mmol/l evaluated by continuous glucose monitoring
Hypoglycaemic events | 16 days
  Beginning of a CGM event is defined as a reading below the threshold for at least 15 min for either a value below 3.0 mmol/l or between 3.9 mmol/l to 3.0 mmol/l. The end of a CGM event is defined as a reading for 15 min above 3.9 mmol/l.

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Herlev Hospital, Copenhagen
  - Rigshospitalet department of endocrinology, Copenhagen
  - Hillerød Hospital, Hillerød
  - Rigshospitalet department of nephrology, København Ø
  - Roskilde Hospital, Roskilde